CLINICAL TRIAL: NCT05662696
Title: Feasibility of Implementing a Mobile Phone-based Telemonitoring Program to Support Pregnant Women at High-risk for Preeclampsia in Karachi, Pakistan
Brief Title: Feasibility of a Telemonitoring Program for Pregnant Women at High-Risk for Preeclampsia in Pakistan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Jinnah Postgraduate Medical Centre (Other Government); Aga Khan University (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-5220
Record Dates: First submitted 2022-10-07; First posted 2022-12-22 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Preeclampsia; Pregnant With Complication
Keywords: Telemonitoring; mHealth; Remote monitoring
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemonitoring Program for Pregnant Women at High Risk for Preeclampsia in Pakistan (Experimental): The study intervention includes a telemonitoring program for high-risk pregnant women, which will be delivered using the telemonitoring platform. The trial will administer the telemonitoring program to 50 pregnant women at high risk for preeclampsia. The intervention will enable pregnant women to take daily blood pressure readings at home with a provided Bluetooth-enabled home blood pressure monitor, to report if participants have symptoms, and to receive automated alerts and self-care messages (e.g., instructing patients to repeat blood pressure readings, call a medical officer, visit the emergency department, etc.). A healthcare provider (medical officer) will receive alerts from the telemonitoring system if the patient's blood pressure trends are out of the target or if the patient is reporting symptoms.
  Interventions: Other: Raabta Telemonitoring Program (Mobile Application)

INTERVENTIONS:
Other: Raabta Telemonitoring Program (Mobile Application) — Raabta is a smartphone application that will allow pregnant women at high-risk for preeclampsia to measure and record daily blood pressure readings and self-reported symptoms. An algorithm is used to generate an alert to a healthcare provider as necessary. The patient also receives an automated alert self-care message based on their measurements and reported symptoms.

SUMMARY:
High maternal mortality from preeclampsia/eclampsia results from a lack of early identification and management of pregnant women at high risk for preeclampsia. A potential tool to support pregnant women at high risk for preeclampsia is telemonitoring. Most telemonitoring interventions have been implemented in high-income countries and thus there is limited evidence on the use and effectiveness of telemonitoring for pregnant women in low-middle-income countries (LMICs). The scarce evidence on the feasibility of telemonitoring program implementation limits the understanding of the process and mechanisms through which the intervention works in LMICs. The study will explore the feasibility of implementing a mobile phone-based telemonitoring program for pregnant women at high-risk for preeclampsia in Karachi, Pakistan. The study will be conducted at the Jinnah Post Graduate Medical Center in Karachi, Pakistan.

The study will use a mixed-methods design to recruit 50 pregnant women at high risk for preeclampsia to assess clinical feasibility across the five foci of Bowen's framework including acceptability, demand, implementation, practicality, and limited-efficacy testing. Data sources will include semi-structured interviews with the patients, and clinicians, as well as data from paper medical records, research logs, and server data. The results of the quantitative and qualitative data will be analyzed separately and then integrated at the interpretation and reporting levels to advance our understanding of the telemonitoring program's feasibility. This will be the first study to provide evidence on the feasibility of using a telemonitoring program where pregnant women at high-risk for preeclampsia in Pakistan will take their own blood pressure readings at home.

DETAILED DESCRIPTION:
Previous studies in LMICs have implemented telemonitoring by community health workers as part of the Community-Level Interventions for Preeclampsia (CLIP) trial and Control of Blood Pressure and Risk Attenuation-Bangladesh, Pakistan, and Sri Lanka [COBRA-BPS] studies. These telemonitoring interventions relied on community health workers to record vital signs on a mobile application during in-person visits, which can miss signs of health issues during physical visits by the community health workers and can also introduce white coat hypertension or masked hypertension. The objective of this study is to enable early risk detection, diagnosis, and treatment of pregnant women at high-risk for preeclampsia between antenatal visits and to provide more frequent data than what can be achieved with home visits by community health workers.

The study intervention will be the telemonitoring program for high-risk pregnant women, which will be delivered using the telemonitoring platform. The telemonitoring program is named "Raabta" which means 'a connection' in Urdu. The Raabta technology has been developed at the Centre for Digital Therapeutics, University Health Network in Toronto, Canada. Hosting of the telemonitoring platform and storage of the patient data will be at the Centre for Digital Therapeutics, University Health Network.

The patient-facing technology includes the Raabta smartphone application (app). The app will enable pregnant women to take daily blood pressure readings at home with a provided Bluetooth-enabled home blood pressure monitor and to receive automated alerts (i.e., self-care messages) via the app. The app will use a rules-based algorithm which is developed using NICE guidelines and consultations from expert clinicians. The algorithm includes settings to trigger alerts and self-care messages for high-risk pregnant women with or without antihypertensives and symptoms of preeclampsia (e.g., instructing patients to repeat blood pressure readings, call a medical officer, visit the emergency department, etc.). Other features of the Raabta app include the use of local language (Urdu), illustrations for daily symptom monitoring questions (for pregnant women who cannot read), an easy-to-understand green-yellow-red alert system that uses the well-known traffic lights analogy, and voice message alerts in conjunction with the text.

The clinician-facing technology includes the web-based Raabta dashboard. To support clinical decision-making, the medical officer situated at the JPMC OB-GYN outpatient department will receive alerts from the telemonitoring system if the patient's blood pressure trends are out of the target or if the patient is reporting symptoms. The medical officer will act as a central point person to communicate with the patients (phone calls or using the asynchronous telemonitoring system chat feature) and with the rest of the participant's care team as needed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at high-risk for preeclampsia (HRPE) who are either in their first or second trimester of pregnancy. The definition of HRPE will follow that of the NICE guidelines that define pregnant women at HRPE as those who have one high-risk factor or more than one moderate risk factor for preeclampsia.
* Participants who can speak and read (at least at a rudimentary level with help from a caregiver) the Urdu language for ease of communication with the research team and to be able to use the telemonitoring system.
* Partners (almost always male husbands in the Pakistani culture) and/or other caregivers (e.g., mother and mother-in-law) of pregnant women [for post-study interviews]
* Clinicians and nurses involved in the implementation of the telemonitoring program [for post-study interviews]

Exclusion Criteria:

* Pregnant women at high-risk for preeclampsia who are admitted to hospital for the management of their preeclampsia condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability | At study completion, approximately 1 year
  Rate of BP Task Compliance for Each Woman (BP readings aimed/sent by women), Rate of Symptom Task Compliance for Each Woman (Symptom readings aimed/sent by women), Compliance of all intended measurements for Each Woman (readings aimed/sent by women) (%), Month-wise Adherence of All Intended Measurements Rate for Each Women (%), Average Overall Adherence Rate of All Intended Measurements for Enrolled Women (%), and Month-wise Overall Adherence Rate of All Intended Measurements for Enrolled Women (%)
Demand | At study completion, approximately 1 year
  Number of Women Consented to Participate in Raabta Program (n), Total Number of Women Enrolled in the Raabta Program (n), Number of Women Decided to Leave the Raabta Program (n), Number of Women Adhered to the Program Until Delivery (n), Length of time each patient enrolled with program/Duration of TM (Weeks), Number of Logins for Each Woman (n), and Total Number of Logins for All Enrolled Women (n)
Practicality | At study completion, approximately 1 year
  Total Number of Calls Made by Medical Officer/Nurse to Each Woman (n), Total Number of Calls Made by Medical Officer/Nurse to All Enrolled Women (n), Total Number of Calls Made by Each Woman to Medical Officer/Nurse (n), Total Number of Calls Made by Enrolled Women (n), Total Number of Emails Received by Medical Officer/Nurse for Alerts (n), Total Number of Request for Changes in Raabta Program (n), and Total Number of Calls Received by Medical Officer/Nurse for Technical Support (n)
Fidelity | At study completion, approximately 1 year
  Total Number of Request for Changes in Raabta Program (n)

SECONDARY OUTCOMES:
Clinical efficacy | At study completion, approximately 1 year
  Presence of PE symptoms (Yes/No), Presence of Gestational Hypertension (Yes/No), Presence of Preeclampsia at Delivery (Yes/No), Presence of Eclampsia at Delivery (Yes/No), Presence of HELLP Syndrome (Yes/No), and Presence of Suspected Fetal Growth Restriction (Yes/No)

OTHER OUTCOMES:
Number of Alerts | At study completion, approximately 1 year
  Total Number of Urgent Alerts (n), Total Number of Non-Urgent Alerts (n), Total Number of Normal Readings (n), Total Number of Red Alerts for Each Woman (n), Total Number of Yellow Alerts for Each Woman (n),
Mean systolic and diastolic blood pressure | At study completion, approximately 1 year
  Mean systolic blood pressure (mmhg), Mean diastolic blood pressure (mmhg)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Seto, PhD, Principal Investigator — University of Toronto

REFERENCES:
- [Derived] Shahil Feroz A, Yasmin H, Saleem S, Bhutta Z, Seto E. Feasibility of implementing a mobile phone-based telemonitoring programme to support pregnant women at high-risk for pre-eclampsia in Karachi, Pakistan: protocol for a mixed-methods study. BMJ Open. 2022 Dec 30;12(12):e070535. doi: 10.1136/bmjopen-2022-070535. PMID 36585144